CLINICAL TRIAL: NCT02018770
Title: Effect of Phototherapy on Pain, Muscles Activity and Joint Mobility in Individuals With Temporomandibular Disorder: A Randomized, Placebo-Controlled and Double-Blind Clinical Trial.
Brief Title: Effect of Phototherapy in Individuals With Temporomandibular Disorder.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Daniela Ap. Biasotto-Gonzalez, Doctor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18032013.4.0000.5511
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-01

CONDITIONS: Temporomandibular Disorder.
Keywords: Temporomandibular Disorders, Electromyogram,; Modalities of physiotherapy,; Temporomandibular dysfunction syndrome,; Lasers.
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phototherapy (Experimental): Three groups will receive different fototerapia of light sources, and group 1 will not receive dose: Group A (0, 65Joules), Group B (1.30 Joules) and Group C (1.95 Joules) .
  Interventions: Radiation: Phototherapy
- Placebo phototherapy (Placebo Comparator): The volunteers will be subjected to the same Groups intervention Phototherapy . The but researcher will receive placebo pen. It is the caveat that, after completed the voluntary participation, will be held with the active pen treatment.
  Interventions: Radiation: Placebo phototherapy

INTERVENTIONS:
Radiation: Phototherapy — Portable Cluster 9 PainAway ® diodes manufactured by Multi Radiance Medical ® (Solon, OH-USA), being 1 905 nm diode (1 mW average power 10 W of peak power, spot of 0.44 cm2), 875 nm diodes 4 (17.5 mW average power for each diode, spot of 1 cm2) and 670 nm diodes 4 (15 mW average power for each diode1 spot, cm2), frequency of 1000 Hz, irradiation time of 300 seconds, energy delivered from 39.3 Joules.
  Arms: Phototherapy
Radiation: Placebo phototherapy — The volunteers will be subjected to the same Groups ' intervention and placebo pen Phototherapy.
  Arms: Placebo phototherapy

SUMMARY:
The present study aims to evaluate the effect of phototherapy with the combination of different sources of light on pain, activity of temporal and masseter muscles, bilateral and joint mobility in subjects with TMD. It will be made a randomized, placebo-controlled and double-blind clinical trial. Individuals participate with myogenic temporomandibular disorder, being allocated into 4 groups randomly and stratified by the method of sealed envelopes. The results will be evaluated using: RDC/TMD, digital caliper, electromyography, and visual analog scale and algometry. The protocols will be used in a single session and will be evaluated in four different moments. The variables that will be investigated are pain, muscle activity and joint mobility. The analyses of the data will be performed by adopting a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years.
* Female volunteers.
* Diagnosis of myogenic TMD pain must masseter presenting moderate to severe according to the RDC / TMD.
* Display body mass index (BMI) less than 25 kg/m2 to standardize the sample.
* In addition, volunteers must submit scores of pain greater than 3 cm according to the Visual Analog Scale masticatory muscles.

Exclusion Criteria:

* history of neurological disorders.
* chronic neck pain resulting from a traumatic incident.
* chronic musculoskeletal condition.
* medical diagnosis of fibromyalgia; systemic disease.
* connective tissue disorder.
* having undergone physical therapy use of analgesic, muscle relaxant.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity. | 1 year
  Will be used a algometry D-200 of Instrutherm ®, which is a semi quantitative method to measure the intensity of the pain by the pressure, find painful spots, in addition to quantify changes the various pain syndromes.

SECONDARY OUTCOMES:
Electromyographic activity | 1 year
  The electrical powers of masticatory muscles will be verified in this study through surface electromyography, specifically the masseter and temporal muscles, serving as a useful tool to quantify muscle activity during Mastication and thus identify its functional changes.

OTHER OUTCOMES:
Analysis of superficial cutaneous temperature | 1 year
  A thermal camera model FLIR T450 ® SC Systems (Stockholm, Sweden) is used to measure the surface skin temperature of the masseter and temporal muscles to verify the effect of phototherapy in them.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ap Biasotto-Gonzalez, Doctor, Principal Investigator — University of Nove de Julho
Locations (1):
- University of Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Herpich CM, Leal-Junior ECP, Gomes CAFP, Gloria IPDS, Amaral AP, Amaral MFRS, Politti F, Biasotto-Gonzalez DA. Immediate and short-term effects of phototherapy on pain, muscle activity, and joint mobility in women with temporomandibular disorder: a randomized, double-blind, placebo-controlled, clinical trial. Disabil Rehabil. 2018 Sep;40(19):2318-2324. doi: 10.1080/09638288.2017.1336648. Epub 2017 Jun 11. PMID 28602137
- [Derived] Herpich CM, Leal-Junior EC, Amaral AP, Tosato Jde P, Gloria IP, Garcia MB, Barbosa BR, El Hage Y, Arruda EE, Gomes CA, Rodrigues MS, de Sousa DF, de Carvalho Pde T, Bussadori SK, Gonzalez Tde O, Politti F, Biasotto-Gonzalez DA. Effects of phototherapy on muscle activity and pain in individuals with temporomandibular disorder: a study protocol for a randomized controlled trial. Trials. 2014 Dec 16;15:491. doi: 10.1186/1745-6215-15-491. PMID 25514875
- See also: URL of the University of Nove de Julho — http://www.uninove.br